CLINICAL TRIAL: NCT03298698
Title: Efficacy of Rituximab in Comparison to Continued Corticosteroid Treatment in Idiopathic Nephrotic Syndrome Unresponsive to 8 Weeks of High Dose Prednisone
Brief Title: Efficacy of Rituximab in Comparison to Continued Corticosteroid Treatment in Idiopathic Nephrotic Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSRNS17
Record Dates: First submitted 2017-08-24; First posted 2017-10-02 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Idiopathic Nephrotic Syndrome; Minimal Change Disease; Focal Segmental Glomerulosclerosis
Keywords: Idiopathic nephrotic syndrome; Minimal change disease; Focal segmental glomerulosclerosis; Rituximab; Randomized clinical trial
MeSH Terms: conditions — Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental | interventions — Rituximab; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab (Experimental): Rituximab: 375 mg/m2 intravenously on day 0 and day 14 B-cells will be monitored weekly, and if no complete depletion is achieved, additional dose(s) of Rituximab will be given at a weekly interval until complete B cell depletion (maximum of 2 additional doses).
  Interventions: Drug: Rituximab
- Prednisone (Active Comparator): Prednisone 1 mg/kg/day (max 80 mg/day) for 8 weeks
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — Rituximab: 375 mg/m2 intravenously on day 0 and day 14 B-cells will be monitored weekly, and if no complete depletion is achieved, additional dose(s) of Rituximab will be given at a weekly interval until complete B cell depletion (maximum of 2 additional doses).
  Other Names: Mabthera
  Arms: Rituximab
Drug: Prednisone — Prednisone 1 mg/kg/day (max 80 mg/day) for 8 weeks
  Other Names: Prednisolone
  Arms: Prednisone

SUMMARY:
This will be an open-label, randomized controlled trial which compares continued treatment with high dose prednisone (standard therapy) to treatment with rituximab in patients with minimal change disease or focal segmental glomerulosclerosis unresponsive to 8 weeks of high dose prednisone .

patients either receive 2 doses of Rituximab 375 mg/m2 iv at time 0 and 14 days with termination of prednisone or standard therapy which consist of 8 additional weeks of high dose prednisone treatment.

DETAILED DESCRIPTION:
Minimal change disease (MCD) and focal segmental glomerulosclerosis (FSGS) are important causes of idiopathic nephrotic syndrome. First-line treatment with high dose prednisone up to 16 weeks is associated with serious side effects. Especially if treatment continues for more than 8 weeks.

Retrospective studies suggested that Rituximab may be more effective in patients unresponsive to 8 weeks of high dose prednisone. Treatment with rituximab was associated with a higher proportion of patients attaining remission of proteinuria and with fewer side effects.

This will be an open-label, randomized controlled trial which compares continued treatment with high dose prednisone (standard therapy) to treatment with rituximab in patients with an idiopathic nephrotic syndrome due to biopsy proven MCD or FSGS age 18 years or older.

All patients will be treated with high dose prednisone (1 mg/kg/day) for 8 weeks.

Patients can be included in the trial in case of persistent persistent proteinuria ≥ 2 g/ 24 hours or a protein-to-creatinine ratio ≥ 2 g/10mmol (2 g/g) after 8 weeks of treatment with high dose prednisone

Patients either receive 2 doses of Rituximab 375 mg/m2 iv at time 0 and 14 days with termination of prednisone or standard therapy which consist of 8 additional weeks of high dose prednisone treatment. In the Rituximab group, B-cells will be monitored weekly, and if no complete depletion is achieved, additional dose(s) of Rituximab will be given at a weekly interval (maximum of 2 additional doses) until complete B cell depletion.

Expected duration of the follow-up is 12 months, consisting of 9 visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Persistent proteinuria ≥ 2 g/ 24 hours or a protein-to-creatinine ratio ≥ 2 g/10mmol (2 g/g) after 8 weeks of treatment with high dose prednisone 1 mg/kg/day (max 80 mg/day)
* Idiopathic nephrotic syndrome caused by biopsy proven minimal change disease or focal segmental glomerulosclerosis

Exclusion Criteria:

* Severe nephrotic syndrome with hypotension
* Previous treatment with immunosuppressive medication other than prednisone
* Treatment with prednisone > 10 weeks in last six months
* Secondary form of FSGS or minimal change disease
* Patients who test positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (anti-HBc).
* Patients infected with HIV or suffering from other active infections
* Patients inoculated with a vaccine within 4 weeks prior to inclusion
* Pregnancy, breast feeding, women with inadequate contraception
* Malignancy
* Kidney transplantation
* Previous treatment with monoclonal antibodies within 2 years prior to inclusion
* Neutrophils < 1.5 x 109/L and/or platelet counts < 75 x 109/L
* Severe heart failure (New York Heart Association Class IV) or severe, uncontrolled cardiac disease
* Active peptic ulcer
* Known hypersensitivity to glucocorticoids
* Insulin resistant diabetes mellitus
* Treatment with carbamazepine, phenobarbital, phenytoin en rifampicin
* Severe osteoporosis with vertebral fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2021-08-22 (Estimated); Study Completion 2022-01-22 (Estimated)

PRIMARY OUTCOMES:
Complete remission | 8 weeks
  The proportion of patients reaching complete remission defined as proteinuria <0.3 g/day or < 300 mg/g

SECONDARY OUTCOMES:
Partial remission | 8 weeks
  The proportion of patients reaching partial remission defined as proteinuria < 3.5 g/24 h or < 3.5 g/g and 50% lower than baseline proteinuria
Late complete or partial remission | 2-12 months
  The proportion of patients reaching complete remission defined as proteinuria <0.3 g/day or < 300 mg/g or The proportion of patients reaching partial remission defined as proteinuria < 3.5 g/24 h or < 3500 mg/g and 50% lower than baseline proteinuria
Time to remission | 12 months
  Time between start of treatment and reaching partial or complete remission
Time to relapse | 12 months
  The time between partial or complete remission and relapse (defined as urinary protein excretion to ≥3.5 g/24 h or ≥3.5 g/g creatinine
Proportion of patients with a relapse | 12 months
  The proportion of patients with relapse (defined as urinary protein excretion to ≥3.5 g/24 h or ≥3.5 g/g creatinine in patients who had at least attained a partial remission and the time to relapse
Proportion of patients treated with additional immunosuppressive drugs | 12 months
  Proportion of patients treated with immunosuppressive drugs other than the assigned treatment with rituximab or prednisolone
General health assessment | at 2, 6, 9 and 12 months
  Difference in general health measured by RAND-36
Quality of life measured with TAAQOL | at 2, 6, 9 and 12 months
  Difference in quality of life measured with TNO-academisch Ziekenhuis Leiden Questionnaire for Adult's Health-Difference in Quality of Life
Proportion of patients with adverse events | at 2 and 12 months
  The proportion of patients with adverse events. Adverse events graded according to Common Terminology Criteria For Adverse Events (NCI-CTCAE v4.03)
Cost-effectiveness analysis | at 2, 6, 9 and 12 months
  Cost-effectiveness will be calculated by dividing the difference in costs by the difference in effectiveness (based on the number of patients in remission) derived from the two groups. The resulting cost-effectiveness ratio will be expressed as costs per one more patient in remission
Cost-utility analysis | at 2, 6, 9 and 12 months
  Cost-utility analysis will be calculated by dividing the difference in costs by the difference in Quality Adjusted Life Years (QALY's). QALY's will be derived from the EuroQol-5d-5L questionnaire.
Difference in kidney function | at 2 and 12 months
  Difference in creatinine clearance and estimated glomerular filtration rate
Proportion of patients with an increase of baseline serum creatinine ≥ 50% | at 2 and 12 months
  The percentage of patients with an increase > 50% of serum creatinine from baseline.
Benefit-risk ratio 1 | at 2 and 12 months
  Difference in the percentage of remissions (benefit) divided by the difference in adverse events grade 3 or 4, including Serious Adverse Events and Suspected Unexpected Serious Adverse Reaction (risk)
Benefit-risk ratio 2 | at 2 and 12 months
  Difference in the percentage of remissions (benefit) divided by the difference in the total number of adverse events (risk)

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen K Deegens, MD,PhD, Principal Investigator — Radboud University Nijmegen Medical center; Jack F Wetzels, MD, PhD, Study Chair — Radboud University Nijmegen Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Azukaitis K, Palmer SC, Strippoli GF, Hodson EM. Interventions for minimal change disease in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2022 Mar 1;3(3):CD001537. doi: 10.1002/14651858.CD001537.pub5. PMID 35230699
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732